CLINICAL TRIAL: NCT06926790
Title: Neoadjuvant Nivolumab Plus Ipilimumab in Resectable Non-small Cell Lung Cancer
Brief Title: Neoadjuvant Nivolumab Plus Ipilimumab in Resectable NSCLC (GALAXY 3)
Acronym: GALAXY 3
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Shuben Li, Director, Training Program of Thoracic Surgery, Director, Section of Tracheal and Pulmonary Surgery, Thoracic Surgery Department, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ES-2025-027-01
Record Dates: First submitted 2025-03-30; First posted 2025-04-15 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancer - Non Small Cell
Keywords: lung cancer; nivolumab plus ipilimumab; neoadjuvant treatment; non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Intervention Model Description: Patients with IIA-IIIB NSCLC received neoadjuvant Nivolumab (3 mg/kg intravenously (i.v.), every 3 week) plus Ipilimumab (1 mg/kg i.v., every 6 week).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Neoadjuvant treatment (Experimental): Patients with IIA-IIIB NSCLC will received 2-3 cycles of neoadjuvant Nivolumab (3 mg/kg intravenously (i.v.), every 3 week) plus Ipilimumab (1 mg/kg i.v., every 6 week).
  Surgery will be performed within 4 to 6 weeks after completion of preoperative therapy.
  After the second cycles treatment, contrast-enhanced chest CT will be performed to evaluate the tumor.
  Interventions: Drug: Nivolumab & Ipilimumab

INTERVENTIONS:
Drug: Nivolumab & Ipilimumab — This study evaluates the safety and efficacy of neoadjuvant nivolumab plus ipilimumab for IIA-IIIB NSCLC. Based on preliminary trial results, this study proposes a new treatment regimen.

SUMMARY:
Neoadjuvant immunotherapy followed by surgery has emerged as the standard treatment for locally advanced and resectable non-small cell lung cancer (NSCLC). However, conventional chemotherapy components may increase treatment-related toxicity, particularly in elderly populations. Additionally, the efficacy of preoperative immunochemotherapy for patients with PD-L1 expression <1% remains to be improved. Emerging evidence has demonstrated that the combination of nivolumab (anti-PD-1) and ipilimumab (anti-CTLA-4) provides superior responses in the treatment of advanced NSCLC. However, the safety and efficacy of this strategy in the neoadjuvant setting remain controversial. Therefore, this single-arm clinical trial aims to evaluate the safety and feasibility of neoadjuvant nivolumab plus ipilimumab followed by surgery in treating locally advanced and resectable NSCLC.

DETAILED DESCRIPTION:
Lung cancer remains the leading cause of cancer-related death globally. Neoadjuvant immunotherapy followed by surgery has been emerged as the standard treatment for locally advanced and resectable non-small cell lung cancer (NSCLC). Numerous clinical trials highlighted the efficacy of preoperative immunochemotherapy, including remarkably shrinking the primary lesion, eliminating micrometastases and ultimately contributing to survival outcomes. Notably, studies also demonstrated neoadjuvant immunochemotherapy increased the access of modified surgery and enhanced survival prognosis of patients with locally advanced NSCLC (IIIB).

Despite these advances, certain limitations remain. Conventional chemotherapy components may elevate treatment-related toxicity, particularly in elderly populations. Additionally, the efficacy of preoperative immunochemotherapy for patients with PD-L1<1% remained to be improve. Emerging evidences demonstrated that nivolumab (anti-PD-1) combine with ipilimumab (antiCTLA-4) provided superior response for the treatment of advanced NSCLC patients. However, the safety and efficacy of this strategy in the neoadjuvant setting remain controversial. Therefore, this single-arm clinical trial aims to evaluate the safety and feasibility of neoadjuvant nivolumab plus ipilimumab followed by surgery in treating locally advanced and resectable NSCLC. The study will enroll 69 eligible participants, with the primary endpoint being pathological complete response (pCR) rate following neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent must be signed.
2. At least 18 years of age.
3. Histologically or cytologically confirmed non-small cell lung cancer (without EGFR, ALK mutation).
4. Have measurable and clinical stage II-IIIA with no known PD-L1 expression or PD-L1 ≤ 1%.
5. disease eligible for surgery.
6. No previous systematic therapy or radiotherapy.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. At least one measurable lesion.
9. No major organ dysfunction, including liver, kidney, and cardiac function.

Exclusion Criteria:

1. Patients with active autoimmune disease or history of autoimmune disease.
2. Patients have received other treatment for non-small cell lung cancer or for any other malignancy.
3. History of allergy to study drug components.
4. Pregnant or breast-feeding.
5. Any mental or psychological condition that would prevent the patient from completing the study or understanding the patient information.
6. Patients who have other malignancies.
7. History of major surgery or serious injury within the past 3 months.
8. HIV, HBV, HCV infection or active pulmonary tuberculosis.
9. Vaccination within 4 weeks prior to the start of the study.
10. Presence of underlying medical conditions that, in the investigator's judgment, could increase the risk associated with study drug administration or interfere with the assessment of toxicity and adverse events.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-10-31 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (PCR) | Within 2 weeks after surgery
  Pathological complete response is predefined as no residual viable tumor cells in primary tumor and lymph nodes.

SECONDARY OUTCOMES:
3-year Event-Free Survival (3-year EFS） | From neoadjuvant treatment to the date of death, recurrence, progression, or the last follow-up (assessed up to 3 years).
  The starting point for EFS was the initiation of neoadjuvant treatment. The endpoint for EFS was defined as the date of death, recurrence, progression, or the last follow-up.
Major Pathological Response (MPR) | Within 2 weeks after surgery
  Major pathological response defined as less than 10% of viable tumor cells in primary tumor.
Safety (Rate of grade 3 and higher grade treatment-related adverse events (TRAEs)) | Between the last dose of neoadjuvant treatment and surgery (assessed up to 30 days)
  Adverse events will be evaluated and recorded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (version 5.0).
Radiological Response | Between the last dose of neoadjuvant treatment and surgery
  Radiographic response will be evaluated according to the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
Postoperative complications | After the surgery assess to 90 days
  Postoperative complications will be evaluated and recorded after the surgery following Clavien-Dindo grade. The minimum and maximum values were grade I-V, and the higher scores mean a worse outcomes.
Intraoperative bleeding | Up to approximately 20 weeks
  Intraoperative bleeding was assessed and recorded by the surgical team. Blood loss was estimated by measuring suction canister volume and weighing surgical sponges, subtracting irrigation fluid.
The Quality of Life | From the Day 1 to at least 90 days after surgery
  The quality of life will be evaluated and recorded according to the EORTC QLQ-C30. The minimum and maximum values were 0-100, and the higher scores mean a better outcome.
Duration of surgery | Up to approximately 20 weeks
  Duration of surgery is the time spent in surgery.
Hospital Stay | Up to approximately 20 weeks
  Hospital Stay is the length of inpatient time spent in hospital.
Feasibility (Completion rate of neoadjuvant treatment and surgery) | From date of treatment allocation until surgery, assessed up to 5 months
  Propotion of patients who complete neoadjuvant treatment and receive surgery within 42 days after neoadjuvant treatment

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Guangzhou Medical University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No